CLINICAL TRIAL: NCT01729845
Title: Mitoxantrone, Etoposide, and Cytarabine (MEC) Following Epigenetic Priming With Decitabine in Adults With Relapsed/Refractory Acute Myeloid Leukemia (AML) or High-Risk Myelodysplastic Syndromes (MDS): A Phase 1/2 Study
Brief Title: Decitabine Followed by Mitoxantrone Hydrochloride, Etoposide, and Cytarabine in Treating Patients With Relapsed or Refractory Acute Myeloid Leukemia or High-Risk Myelodysplastic Syndromes
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Fred Hutchinson Cancer Center (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Principal Investigator, Anna Halpern, Principal Investigator, Fred Hutchinson Cancer Center
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2652.00; NCI-2012-02224 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); 2652; FH#2652; 2652.00 (Other: Fred Hutch/University of Washington Cancer Consortium); P30CA015704 (NIH)
Record Dates: First submitted 2012-11-15; First posted 2012-11-20 (Estimated); Results first posted 2018-01-12 (Actual); Last update posted 2019-02-07 (Actual); Status verified 2019-02

CONDITIONS: Previously Treated Myelodysplastic Syndrome; Recurrent Adult Acute Myeloid Leukemia
MeSH Terms: conditions — Leukemia, Myeloid, Acute | interventions — Cytarabine; Decitabine; Injections; Etoposide; Mitoxantrone

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Treatment (decitabine, MEC) (Experimental): Patients receive decitabine IV on days -9 to -5 (dose level 1), days -11 to -5 (dose level 2), or days -14 to -5 (dose level 3).
  INDUCTION THERAPY: Patients receive mitoxantrone hydrochloride IV on days 1-5, etoposide IV on days 1-5, and cytarabine IV on days 1-5. Patients achieving CR or CR with CRp may receive up to 2 courses of induction therapy and up to 2 courses of consolidation therapy.
  Interventions: Drug: Cytarabine; Drug: Decitabine; Drug: Etoposide; Other: Laboratory Biomarker Analysis; Drug: Mitoxantrone Hydrochloride

INTERVENTIONS:
Drug: Cytarabine — Given IV
  Other Names: .beta.-Cytosine arabinoside; 1-.beta.-D-Arabinofuranosyl-4-amino-2(1H)pyrimidinone; 1-.beta.-D-Arabinofuranosylcytosine; 1-Beta-D-arabinofuranosyl-4-amino-2(1H)pyrimidinone; 1-Beta-D-arabinofuranosylcytosine; 1.beta.-D-Arabinofuranosylcytosine; 2(1H)-Pyrimidinone, 4-Amino-1-beta-D-arabinofuranosyl-; 2(1H)-Pyrimidinone, 4-amino-1.beta.-D-arabinofuranosyl-; Alexan; Ara-C; ARA-cell; Arabine; Arabinofuranosylcytosine; Arabinosylcytosine; Aracytidine; Aracytin; Aracytine; Beta-Cytosine Arabinoside; CHX-3311; Cytarabinum; Cytarbel; Cytosar; Cytosar-U; Cytosine Arabinoside; Cytosine-.beta.-arabinoside; Cytosine-beta-arabinoside; Erpalfa; Starasid; Tarabine PFS; U 19920; U-19920; Udicil; WR-28453
Drug: Decitabine — Given IV
  Other Names: 5-Aza-2'-deoxycytidine; Dacogen; Decitabine for Injection; Deoxyazacytidine; Dezocitidine
Drug: Etoposide — Given IV
  Other Names: Demethyl Epipodophyllotoxin Ethylidine Glucoside; EPEG; Lastet; Toposar; Vepesid; VP 16-213; VP-16; VP-16-213
Other: Laboratory Biomarker Analysis — Correlative studies
Drug: Mitoxantrone Hydrochloride — Given IV
  Other Names: CL 232315; DHAD; DHAQ; Dihydroxyanthracenedione Dihydrochloride; Mitoxantrone Dihydrochloride; Mitoxantroni Hydrochloridum; Mitozantrone Hydrochloride; Mitroxone; Neotalem; Novantrone; Onkotrone; Pralifan

SUMMARY:
This phase I/II trial studies the side effects and best dose of decitabine followed by mitoxantrone hydrochloride, etoposide, and cytarabine and to see how well they work in treating patients with acute myeloid leukemia or high-risk myelodysplastic syndrome that has returned after a period of improvement or does not respond to treatment. Drugs used in chemotherapy, such as mitoxantrone hydrochloride, etoposide, cytarabine, and decitabine, work in different ways to stop the growth of cancer cells, either by killing the cells, by stopping them from dividing, or by stopping them from spreading. Giving more than one drug (combination chemotherapy) may kill more cancer cells.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. Estimate the maximum tolerated dose (MTD) of decitabine priming followed by sequential mitoxantrone hydrochloride/etoposide/cytarabine (MEC) chemotherapy in adults with relapsed/refractory acute myeloid leukemia (AML).

SECONDARY OBJECTIVES:

I. Determine, within the limits of a Phase 1/2 study, disease response and duration of remission.

II. Identify biomarkers (e.g., deoxyribonucleic acid [DNA] methylation and/or gene expression changes) associated with treatment responses.

OUTLINE: This is a phase I, dose-escalation study of decitabine followed by a phase II study.

Patients receive decitabine intravenously (IV) on days -9 to -5 (dose level 1), days -11 to -5 (dose level 2), or days -14 to -5 (dose level 3).

INDUCTION THERAPY: Patients receive mitoxantrone hydrochloride IV on days 1-5, etoposide IV on days 1-5, and cytarabine IV on days 1-5. Patients achieving complete response (CR) or CR with incomplete platelet count recovery (CRp) may receive up to 2 courses of induction therapy and up to 2 courses of consolidation therapy.

After completion of study treatment, patients are followed up every 3 months for up to 5 years.

ELIGIBILITY:
Inclusion Criteria:

* Prior diagnosis of "high-risk" myelodysplastic syndrome (MDS) (>= 10% blasts) or AML other than acute promyelocytic leukemia (APL) with t(15;17) (q22;q12) or variants according to the 2008 World Health Organization (WHO) classification; patients with biphenotypic AML are eligible
* Relapsed/persistent disease according to standard criteria requiring salvage therapy; outside diagnostic material is acceptable as long as peripheral blood and/or bone marrow slides are reviewed at the study institution; flow cytometric analysis of peripheral blood and/or bone marrow should be performed according to institutional practice guidelines
* Patients with prior autologous or allogeneic hematopoietic cell transplantation (HCT) are eligible if relapse occurs provided symptoms of graft-versus host disease are well controlled with stable use of immunosuppressive agents
* Treatment-related mortality (TRM) score =< 9.2 as calculated with simplified model
* Should be off any active therapy for AML with the exception of hydroxyurea for at least 14 days prior to study registration unless patient has rapidly progressive disease, and all grade 2-4 non-hematologic toxicities should have resolved
* May have previously received monotherapy with demethylating agents for MDS or AML
* May have previously received chemotherapy with MEC for MDS or AML
* Patients with symptoms/signs of hyperleukocytosis or white blood cells (WBC) > 100,000/uL can be treated with leukapheresis or may receive up to 2 doses of cytarabine (up to 500 mg/m^2/dose) prior to enrollment
* Bilirubin =< 2 x institutional upper limit of normal (IULN) unless elevation is thought to be due to hepatic infiltration by AML, Gilbert's syndrome, or hemolysis (assessed within 7 days prior to study day 1)
* Serum creatinine =< 1.5 x IULN (assessed within 7 days prior to study day 1)
* Left ventricular ejection fraction >= 40%, assessed within 3 months prior to study day 1, e.g. by multi gated acquisition (MUGA) scan or echocardiography, or other appropriate diagnostic modality and no clinical evidence of congestive heart failure; if the patient had anthracycline-based therapy since the most recent cardiac assessment, cardiac evaluation should be repeated if there is clinical or radiographical suspicion of cardiac dysfunction, or if the previous cardiac assessment was abnormal
* Women of childbearing potential and men must agree to use adequate contraception
* Provide written informed consent

Exclusion Criteria:

* Refractory/relapsing myeloid blast crisis of chronic myeloid leukemia (CML), unless patient is not considered candidate for tyrosine kinase inhibitor treatment
* Concomitant illness associated with a likely survival of < 1 year
* Active systemic fungal, bacterial, viral, or other infection, unless disease is under treatment with anti-microbials and/or controlled or stable (e.g. if specific, effective therapy is not available/feasible or desired [e.g. chronic viral hepatitis, human immunodeficiency virus (HIV)]); patient needs to be clinically stable as defined as being afebrile and hemodynamically stable for 24 hours; patients with fever thought to be likely secondary to leukemia are eligible
* Known hypersensitivity to any study drug
* Pregnancy or lactation
* Patients may not be receiving any other investigational agents

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 52 (Actual)
Dates: Start 2012-12-20 (Actual); Primary Completion 2016-08-25 (Actual); Study Completion 2017-04-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Anna Halpern, Principal Investigator — Fred Hutch/University of Washington Cancer Consortium
Locations (3):
- United States (3):
  - Kadlec Clinic Hematology and Oncology, Kennewick, Washington
  - EvergreenHealth Medical Center, Kirkland, Washington
  - Fred Hutch/University of Washington Cancer Consortium, Seattle, Washington

RESULTS

PARTICIPANT FLOW:
Groups:
- Dose Level 1: 5-Days of Decitabine-MEC: Patients receive decitabine IV days -9 to -5 (dose level 1).
  INDUCTION THERAPY: Patients receive mitoxantrone hydrochloride IV on days 1-5, etoposide IV on days 1-5, and cytarabine IV on days 1-5. Patients achieving CR or CR with CRp may receive up to 2 courses of induction therapy and up to 2 courses of consolidation therapy.
  Cytarabine: Given IV
  Decitabine: Given IV
  Etoposide: Given IV
  Mitoxantrone Hydrochloride: Given IV
- Dose Level 2: 7-Days of Decitabine-MEC: Patients receive decitabine IV days -11 to -5 (dose level 2).
  INDUCTION THERAPY: Patients receive mitoxantrone hydrochloride IV on days 1-5, etoposide IV on days 1-5, and cytarabine IV on days 1-5. Patients achieving CR or CR with CRp may receive up to 2 courses of induction therapy and up to 2 courses of consolidation therapy.
  Cytarabine: Given IV
  Decitabine: Given IV
  Etoposide: Given IV
  Mitoxantrone Hydrochloride: Given IV
- Dose Level 3: 10-days of Decitabine-MEC: Patients receive decitabine IV days -14 to -5 (dose level 3).
  INDUCTION THERAPY: Patients receive mitoxantrone hydrochloride IV on days 1-5, etoposide IV on days 1-5, and cytarabine IV on days 1-5. Patients achieving CR or CR with CRp may receive up to 2 courses of induction therapy and up to 2 courses of consolidation therapy.
  Cytarabine: Given IV Decitabine: Given IV Etoposide: Given IV Mitoxantrone Hydrochloride: Given IV
Period: Safety/Tolerability of Dec/MEC
Arm/Group | Dose Level 1: 5-Days of Decitabine-MEC | Dose Level 2: 7-Days of Decitabine-MEC | Dose Level 3: 10-days of Decitabine-MEC
Started | 6 | 34 | 12
Completed | 6 | 34 | 12
Not Completed | 0 | 0 | 0
Period: Efficacy of Dec/MEC
Arm/Group | Dose Level 1: 5-Days of Decitabine-MEC | Dose Level 2: 7-Days of Decitabine-MEC | Dose Level 3: 10-days of Decitabine-MEC
Started | 0 | 22 | 0
Completed | 0 | 22 | 0
Not Completed | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Dose Level 1: 5-Days of Decitabine-MEC: Patients receive decitabine IV days -9 to -5 (dose level 1).
  INDUCTION THERAPY: Patients receive mitoxantrone hydrochloride IV on days 1-5, etoposide IV on days 1-5, and cytarabine IV on days 1-5. Patients achieving CR or CR with CRp may receive up to 2 courses of induction therapy and up to 2 courses of consolidation therapy.
  Cytarabine: Given IV
  Decitabine: Given IV
  Etoposide: Given IV
  Laboratory Biomarker Analysis: Correlative studies
  Mitoxantrone Hydrochloride: Given IV
- Dose Level 2: 7-Days of Decitabine-MEC: Patients receive decitabine IV days -11 to -5 (dose level 2).
  INDUCTION THERAPY: Patients receive mitoxantrone hydrochloride IV on days 1-5, etoposide IV on days 1-5, and cytarabine IV on days 1-5. Patients achieving CR or CR with CRp may receive up to 2 courses of induction therapy and up to 2 courses of consolidation therapy.
  Cytarabine: Given IV
  Decitabine: Given IV
  Etoposide: Given IV
  Laboratory Biomarker Analysis: Correlative studies
  Mitoxantrone Hydrochloride: Given IV
- Dose Level 3: 10-Days of Decitabine-MEC: Patients receive decitabine IV days -14 to -5 (dose level 3).
  INDUCTION THERAPY: Patients receive mitoxantrone hydrochloride IV on days 1-5, etoposide IV on days 1-5, and cytarabine IV on days 1-5. Patients achieving CR or CR with CRp may receive up to 2 courses of induction therapy and up to 2 courses of consolidation therapy.
  Cytarabine: Given IV
  Decitabine: Given IV
  Etoposide: Given IV
  Laboratory Biomarker Analysis: Correlative studies
  Mitoxantrone Hydrochloride: Given IV
- Total: Total of all reporting groups
Arm/Group | Dose Level 1: 5-Days of Decitabine-MEC | Dose Level 2: 7-Days of Decitabine-MEC | Dose Level 3: 10-Days of Decitabine-MEC | Total
Number analyzed (Participants) | 6 | 34 | 12 | 52
Age, Continuous [Median (Full Range); unit: years] | 54 [54 to 66] | 55 [19 to 70] | 57 [32 to 72] | 55 [19 to 72]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 1 | 16 | 6 | 23
  Male | 5 | 18 | 6 | 29

OUTCOME MEASURES:

1. Primary Outcome: Most Efficacious and Tolerated Dosage of Decitabine (Period 1)
Description: MTD (most tolerated dose) of decitabine, measured in number of dose limiting toxicities. MTD defined as the highest dose in which the incidence of dose limiting toxicity is < 33%, graded according to the National Cancer Institute Common Terminology Criteria for Adverse Events version 4.0 (Phase I)
Time Frame: through day 45
Measure: Number; unit: Incidents
Groups:
- Dose Level 1: 5-Days of Decitabine-MEC: Patients receive decitabine IV days -9 to -5 (dose level 1). INDUCTION THERAPY: Patients receive mitoxantrone hydrochloride IV on days 1-5, etoposide IV on days 1-5, and cytarabine IV on days 1-5. Patients achieving CR or CR with CRp may receive up to 2 courses of induction therapy and up to 2 courses of consolidation therapy.
  Cytarabine: Given IV Decitabine: Given IV Etoposide: Given IV Laboratory Biomarker Analysis: Correlative studies Mitoxantrone Hydrochloride: Given IV
  Decitabine: Given IV
  Etoposide: Given IV
  Mitoxantrone Hydrochloride: Given IV
- Dose Level 3: 10-Days of Decitabine-MEC: Patients receive decitabine IV days -14 to -5 (dose level 1).
  INDUCTION THERAPY: Patients receive mitoxantrone hydrochloride IV on days 1-5, etoposide IV on days 1-5, and cytarabine IV on days 1-5. Patients achieving CR or CR with CRp may receive up to 2 courses of induction therapy and up to 2 courses of consolidation therapy.
  Cytarabine: Given IV Decitabine: Given IV Etoposide: Given IV Laboratory Biomarker Analysis: Correlative studies Mitoxantrone Hydrochloride: Given IV
Arm/Group | Dose Level 1: 5-Days of Decitabine-MEC | Dose Level 2: 7-Days of Decitabine-MEC | Dose Level 3: 10-Days of Decitabine-MEC
Number analyzed (Participants) | 6 | 12 | 12
Incidents
  Dose-limiting toxiticies | 0 | 0 | 0
  Complete Remission | 1 | 5 | 3
  Complete Remission, incomplete PLT recovery | 2 | 1 | 2
  Complete Remission, incomplete blood count recover | 0 | 1 | 0
  Morphologic leukemia-free state | 0 | 0 | 3
  Resistant Disease | 1 | 3 | 4
  Death (among those who received MEC) | 2 | 1 | 0

2. Secondary Outcome: Remission Rate Including CR and CRp
Description: Complete remission (CR) and Complete remission with incomplete platelet recovery (CRp) categorized according to criteria recommended by International Working Groups:
  Complete resolution of disease-related symptoms and signs including palpable hepatosplenomegaly; hemoglobin level at least 110 g/L, platelet count at least 100x10^9/L, and absolute neutrophil count at least 1.0 x10^9/L. In addition, all 3 blood counts should be no higher than the upper normal limit; Normal leukocyte differential; Bone marrow histologic remission defined as the presence of age-adjusted normocellularity, no more than 5% myeloblasts, and an osteomyelofibrosis grade no higher than 1.
Time Frame: Up to 5 years
Population: Population includes all Dose Level 2 participants from both periods 1 and 2.
Measure: Count of Participants; unit: Participants
Arm/Group | Dose Level 2: 7-Days of Decitabine-MEC
Number analyzed (Participants) | 34
Participants | 11

3. Secondary Outcome: Duration of Relapse-free Survival (for Patients Achieving CR or CRp)
Description: Categorized according to criteria recommended by International Working Groups.
Time Frame: Up to 5 years
Population: Population includes all Dose Level 2 participants, from both periods 1 and 2, who achieved CR or CRp
Measure: Median (Full Range); unit: Days
Groups:
- Dose Level 2: 7-Days of Decitabine-MEC: Patients receive decitabine IV on days -11 to -5 (dose level 2)
  INDUCTION THERAPY: Patients receive mitoxantrone hydrochloride IV on days 1-5, etoposide IV on days 1-5, and cytarabine IV on days 1-5. Patients achieving CR or CR with CRp may receive up to 2 courses of induction therapy and up to 2 courses of consolidation therapy.
  Cytarabine: Given IV
  Decitabine: Given IV
  Etoposide: Given IV
  Mitoxantrone Hydrochloride: Given IV
Arm/Group | Dose Level 2: 7-Days of Decitabine-MEC
Number analyzed (Participants) | 11
Days | 150 [20 to 1031]

4. Secondary Outcome: Overall Survival
Description: Survival measured as of day of last contact. Categorized according to criteria recommended by International Working Groups.
Time Frame: Up to 5 years
Population: Population includes all Dose Level 2 participants, from both periods 1 and 2.
Measure: Median (Full Range); unit: days
Arm/Group | Dose Level 2: 7-Days of Decitabine-MEC
Number analyzed (Participants) | 34
days | 564 [165 to 1239]

ADVERSE EVENTS:
Description: Death's reported were not reportable Serous adverse events per protocol. They were expected, or not related to drug and/or described in the protocol and consent form.
Arm/Group | Dose Level 1: 5-Days of Decitabine-MEC | Dose Level 2: 7-Days of Decitabine-MEC | Dose Level 3: 10-days of Decitabine-MEC
All-Cause Mortality (participants affected / at risk) | 2/6 | 1/34 | 0/12
Serious Adverse Events (participants affected / at risk) | 0/6 | 0/34 | 0/12
Other Adverse Events (participants affected / at risk) | 6/6 | 33/34 | 12/12
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Dose Level 1: 5-Days of Decitabine-MEC (N=6) | Dose Level 2: 7-Days of Decitabine-MEC (N=34) | Dose Level 3: 10-days of Decitabine-MEC (N=12)
Febrile Neutropenia (Blood and lymphatic system disorders) | 5 | 27 | 11
Maculopapular Rash (Skin and subcutaneous tissue disorders) | 1 | 1 | 1
Sepsis (Infections and infestations) | 1 | 10 | 5
Bacteremia (Infections and infestations) | 1 | 12 | 5
Pneumonia (Infections and infestations) | 1 | 1 | 1
Fungal Pneumonia (Infections and infestations) | 1 | 8 | 4
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 1 | 5 | 4
Respitatory Failure (Respiratory, thoracic and mediastinal disorders) | 1 | 5 | 3
Respiratory Tract infection (Infections and infestations) | 2 | 0 | 1
Diarrhea (Gastrointestinal disorders) | 0 | 2 | 2
Anorexia (Metabolism and nutrition disorders) | 0 | 2 | 2
Mucositis (Respiratory, thoracic and mediastinal disorders) | 1 | 12 | 0
C Diff (Gastrointestinal disorders) | 0 | 2 | 2
Hypokalemia (Metabolism and nutrition disorders) | 0 | 2 | 2
Hyponatremia (Metabolism and nutrition disorders) | 2 | 1 | 3
Syncope (Nervous system disorders) | 0 | 2 | 0
Soft Tissue Infection (Infections and infestations) | 0 | 4 | 0
Sinusitis (Infections and infestations) | 0 | 3 | 0
Nausea (Gastrointestinal disorders) | 1 | 3 | 1
Esophagitis (Gastrointestinal disorders) | 0 | 4 | 0
Atrial Tachycardia (Cardiac disorders) | 1 | 0 | 0
Hypotension (Vascular disorders) | 0 | 2 | 0
Tropinemia/NSTEMI (Cardiac disorders) | 0 | 2 | 0
Tumor Lysis (Metabolism and nutrition disorders) | 0 | 1 | 1
Colitis (Gastrointestinal disorders) | 0 | 0 | 1
Elevated BR (Respiratory, thoracic and mediastinal disorders) | 0 | 2 | 0
Edema limbs (General disorders) | 0 | 0 | 1
Cholecystitis (Gastrointestinal disorders) | 0 | 2 | 0
Enteritis (Gastrointestinal disorders) | 0 | 0 | 1
Vomiting (Gastrointestinal disorders) | 0 | 3 | 1
Pulmonary Embolism (Vascular disorders) | 0 | 2 | 1
Anxiety (Psychiatric disorders) | 0 | 1 | 1
Acute Kidney Injury (Renal and urinary disorders) | 0 | 2 | 1
Elevated Liver Function Tests (Investigations) | 0 | 1 | 2
Hypophosphatemia (Metabolism and nutrition disorders) | 0 | 2 | 1
Hypocalcemia (Metabolism and nutrition disorders) | 0 | 0 | 1
Catheter Infection (Infections and infestations) | 0 | 2 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes